CLINICAL TRIAL: NCT01855061
Title: Feasibility Study of Biomarker Development for Response Prediction by Large Scale DNA Mutational Analysis of Metastatic Lesions
Brief Title: Biomarker Development for Response Prediction by DNA Mutational Analysis
Acronym: CPCT-01
Status: Terminated | Type: Observational
Sponsor: P.O. Witteveen (Other)
Collaborators: Erasmus Medical Center (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, P.O. Witteveen, Investigator, UMC Utrecht
Organization: UMC Utrecht (Other)
Other Study IDs: NL35198.041.11
Record Dates: First submitted 2011-08-01; First posted 2013-05-16 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Neoplasm Metastasis
Keywords: Feasibility studies; Sequence analysis, DNA; Biological markers; Solid tumors; Neoplasm metastasis; Irinotecan; Pharmacokinetics SN-38; Carboxylesterase activity within metastasis
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Blood Specimen Collection; Pharmacokinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Histological biopsies Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Irinotecan: Patients will be subjected to a their metastatic solid tumor. Radiological response will be evaluated after each 2 cycles: 1. percentage change in radiological volume of the "index lesion" (radiological measurable lesion that underwent biopsy) after the first two cycles of irinotecan; 2. radiological response according to RECIST 1.1 after each 2 cycles. Patients are intended to receive irinotecan until progressive disease or unacceptable toxicity. Patients will be subjected to another biopsy of the index lesion at definitive discontinuation of irinotecan. Patients will also be subjected to blood draws for determining patient's genetic background variation.
  Side studies include:
  * pharmacogenetics
  * pharmacokinetics of SN-38
  * carboxylesterase activity in the index lesion
  * midazolam clearance test (only in Rotterdam patients)
  Interventions: Procedure: Biopsy; Procedure: Blood samples; Procedure: Pharmacokinetics; Procedure: Midazolam clearance test

INTERVENTIONS:
Procedure: Biopsy — Histological biopsy of the "index lesion" (a radiological measurable lesion on which biopsy is performed) at baseline, as well as when showing progressive disease. Histological biopsies will be subjected to DNA sequencing to assess the mutational profile, as well as to analysis of carboxylesterase activity.
  Other Names: Histological biopsy
Procedure: Blood samples — Blood samples will be taken at baseline to determine patient's genetic background variation (germline DNA).
  Other Names: Blood sampling
Procedure: Pharmacokinetics — Blood samples will be taken for pharmacokinetic analysis of the active irinotecan metabolite (SN-38).
  Other Names: PK; Pharmacokinetic analysis; Pharmacokinetic analyses
Procedure: Midazolam clearance test — Patients who are being treated in Rotterdam will be subjected to blood draws for validation of the earlier developed midazolam phenotyping test (midazolam clearance test), which may be an indicator for pharmacokinetics of irinotecan.
  Other Names: MCT

SUMMARY:
The purpose of this study is to determine whether it is possible to predict response to chemotherapy in patients with metastatic cancer who are treated with irinotecan by determining the mutational profile of the tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a metastatic solid tumor who have failed at least one line of palliative chemotherapy and are irinotecan naïve.
2. Patients who are, as per local protocol, eligible for palliative treatment with (standard of care) irinotecan.
3. Measurable metastatic lesion(s), according to RECIST 1.1 criteria.
4. Radiological measurable metastatic lesion(s) of which a histological biopsy can safely be obtained:

   1. Patients with safely accessible metastases.
   2. Patients not known with bleeding disorders (such as hemophilia) or bleeding complications from biopsies, dental procedures or surgeries.
   3. Patients not using any anti-coagulant medication at the time of biopsy: all aspirin derivatives, NSAID's, coumarines, platelet function inhibitors, heparins (including LMWHs) and oral factor Xa inhibitors are not allowed, unless medication can either be safely stopped or counteracted.
   4. Adequate coagulation status on the day of biopsy as measured by:

      * PTT < 1.5 x ULN
      * APTT < 1.5 x ULN
      * Platelet count 100 x 10*9 / L or higher
      * PT-INR < 1.6
      * HB > 6
   5. Biopsies should be performed at least four weeks after last bevacizumab administration.
5. Patients age 18 years or up, willing and able to comply with the protocol as judged by the investigator with a signed informed consent.

Exclusion Criteria:

Patients not meeting all of the above inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a metastatic solid tumor who are eligible for (standard of care) treatment with irinotecan.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2011-05; Primary Completion 2015-11 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Exploration of the correlation between the mutational profile and the percentage change in volumetric measurement of the index lesion after the first two cycles of chemotherapy. | Change in radiological volume of the index lesion after the first 2 cycles of irinotecan. Radiological response (according to RECIST 1.1) after the first 2 cycles of irinotecan (i.e. after 2 x 3 weeks = 6 weeks)

SECONDARY OUTCOMES:
Exploration of the correlation between the mutational profile and radiological response according to RECIST-criteria after the first two cycles of chemotherapy. | Analysis 6 weeks after initiation of treatment
Exploration of the correlation between the mutational profile and progression free survival and overall survival. | Overall survival approximately after 2 years of first cycle of irinotecan. Progression free survival approximately 3 months after first irinotecan
Exploration of the correlation between the mutational profile of the index lesion and patient's germline DNA background variation. | Analysis after progressive disease, on average after 3 months.
Differences in mutational profile of metastasis prior to and after exposure to treatment. | Analysis after progressive disease and subsequent post-treatment biopsy, on average after 3 months of treatment
Determine reliable and valid strategies for statistical analysis for biomarker discovery | 2 years
Correlate response to pharmacokinetics of SN-38 | After progressive disease and subsequent post-treatment biopsy, in general after 3 months of treatment
Determine carboxylesterase activity in metastatic tumor material (pre- and posttreatment) and correlate intra-tumoral carboxylesterase activity to systemic SN-38 pharmacokinetics and to irinotecan response | After progressive disease and subsequent post-treatment biopsy, in general after 3 months of treatment
Determine clinical applicability of the midazolam phenotyping probe | After first cycle of irinotecan, at three weeks
Number and nature of all (serious) adverse events of study related procedures | 14 days after baseline biopsy and 14 days after post-treatment biopsy (approximately after 3 months of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Langenberg, MD/PhD, Principal Investigator — UMC Utrecht; Neeltje Steeghs, MD/PhD, Principal Investigator — Netherlands Cancer Institute - Antoni van Leeuwenhoek hospital, Amsterdam; Ron Mathijssen, MD/PhD, Principal Investigator — Erasmus Medical Center - Daniël den Hoed clinic, Rotterdam
Locations (3):
- Netherlands (3):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, North Holland
  - Erasmsus Medical Center - Daniël den Hoed clinic, Rotterdam, South Holland
  - University Medical Center Utrecht, Utrecht